CLINICAL TRIAL: NCT01138709
Title: Phase II Vitala 12 Hour Wear Test With Convex Products
Brief Title: Vitala 12 Hour Wear Test With Convex Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CC-0196-09-A721
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2013-07

CONDITIONS: End Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Convexity/Vitala (Experimental): For all enrolled Subjects, STAGE 1 (Days 1 - 14 equals Convex Product Wear Period followed by, for those who successfully complete Stage I, weekly increases in wear time of the Vitala™ device beginning with 4 hours of daily wear per week (Days 15 to 21), followed by 8 hours of daily wear time per week (Day 22 to 28), followed by 12 hours of daily wear time (Days 29 to 43).
  Interventions: Device: Vitala

INTERVENTIONS:
Device: Vitala — Vitala™ Continence Control Device

SUMMARY:
The primary objective of this phase II clinical trial is to assess the safety of the Vitala™ device during 12 hours of daily wear with convex products.

ELIGIBILITY:
Inclusion Criteria:

* Is of legal consenting age.
* Is able to read, write, and understand the study, the required procedures, and the study related documentation.
* Has signed the informed consent.
* Has an end colostomy of at least 12 weeks duration with formed or semi-formed effluent.
* Currently uses a convex skin barrier wafer or uses convex inserts into standard skin barrier wafers or is willing to wear SUR-FIT Natura® Durahesive® Skin Barrier with CONVEX-IT® or SUR-FIT Natura® Disposable Convex Inserts in 45mm or 57mm flange sizes. Enrollment will target 15 current convex product users and 10 non convex users.
* The investigator is relatively sure the subject will be able to wear a SUR-FIT Natura® Durahesive® Skin Barrier with CONVEX-IT® in 45mm or 57mm flange size with a stoma opening size from 13mm up to 50mm or the SUR-FIT Natura® Disposable Convex Inserts in 45mm or 57mm flange sizes.
* Is willing to remove and replace the skin barrier wafer after three days, more often if desired, during Stage 2.
* Has a stoma that protrudes no more than 2 cm at rest (lying down on back).
* Has demonstrated success in wearing a traditional pouching system. (Investigator judgment)
* Is willing to participate in the trial for a total of 43 days.
* Is willing to meet with the investigator for a total of 5 scheduled visits plus additional visits as deemed necessary by the investigator.
* Has the ability to do complete self-care.

Exclusion Criteria:

* Has known skin sensitivity to any component of the products being tested.
* Has a skin rating of "2" or greater according to the Skin Rating Scale.
* Has peristomal ulcerations, peristomal pressure necrosis, parastomal hernia, Caput Medusa or mucocutaneous separation.
* Is receiving radiation in the area of the pouching system.
* Is receiving chemotherapy other than a stable regimen of maintenance chemotherapy.
* Requires a pouch belt while wearing Vitala™.
* Requires a moldable skin barrier.
* Has participated in a clinical study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Assessment of safety during 12 hours of Vitala™ device wear with convex products by measuring the frequency of adverse events relating to the stoma (including gastrointestinal, stomal and surrounding skin events), and stomal vascularity. | 29 Days
  Assess safety during 12 hours of Vitala™ device wear with convex products by measuring the frequency of adverse events relating to the stoma (including gastrointestinal, stomal and surrounding skin events), and stomal vascularity.
Assessment of the Efficacy in the Restoration of Continence (absence of fecal leakage around the device) for 29 days of Vitala™ daily wear according to the following parameters. | 29 Days
  Restoration of Continence (absence of fecal leakage around the device) for 29 days of Vitala™ daily wear according to the following parameters:
  * Proportion of subjects with leakage over time.
  * Overall weighted leakage rate.
  * Proportion of subjects without leakage.
  * Self-rating of ability to restore continence.

SECONDARY OUTCOMES:
Assessment of the Efficacy of Vitala™ device will also be evaluated for the following efficacy parameters. | 29 Days
  Vitala™ device will also be evaluated for the following efficacy parameters:
  * Security of the device.
  * Flange to flange security.
  * Device wear time.
  * Subject comfort.
  * Control of odor.
  * Control of noise due to flatus release from the stoma.
  * Ease of use of the device during application and removal.
  * Subject acceptance of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Dheerendra Kommala, MD, Study Director — ConvaTec Inc.
Locations (5):
- United States (5):
  - Non-Institutional Investigator, Tucson, Arizona
  - ET Nursing Services, Jacksonville, Florida
  - Restored Images, Kansas City, Missouri
  - Image Specialties, Saint Joseph, Missouri
  - Non-Institutional Investigator, Reynoldsburg, Ohio